CLINICAL TRIAL: NCT01810874
Title: STELLA Trial: Staging of Endometrial and Ovarian Cancer Comparing the Transperitoneal vs. Extraperitoneal Approach for Laparoscopic Lymphadenectomy of Aortic Nodes
Brief Title: STELLA Trial: Transperitoneal vs. Extraperitoneal Approach for Laparoscopic Staging of Endometrial/Ovarian Cancer
Acronym: STELLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Fundación Mutua Madrileña (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: STELLA
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Endometrial Neoplasms; Ovarian Neoplasms
Keywords: extraperitoneal; transperitoneal; laparoscopic aortic lymphadenectomy; endometrial ovarian cancer; ovarian cancer; surgical staging
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transperitoneal (Active Comparator): Patients who where randomized to transperitoneal laparoscopic aortic lymphadenectomy.
  Interventions: Procedure: Transperitoneal laparoscopic aortic lymphadenectomy
- Extraperitoneal (Experimental): Patients who where randomized to extraperitoneal laparoscopic aortic lymphadenectomy.
  Interventions: Procedure: Extraperitoneal laparoscopic aortic lymphadenectomy

INTERVENTIONS:
Procedure: Transperitoneal laparoscopic aortic lymphadenectomy — Aortic/para-aortic lymph nodes dissection and retrieval by transperitoneal laparoscopy; the intervention may be completed by robotic-assisted or traditional laparoscopy.
  Other Names: Transperitoneal laparoscopic para-aortic lymphadenectomy
  Arms: Transperitoneal
Procedure: Extraperitoneal laparoscopic aortic lymphadenectomy — Aortic/para-aortic lymph nodes dissection and retrieval by extraperitoneal laparoscopy; the intervention may be completed by robotic-assisted or traditional laparoscopy.
  Other Names: Extraperitoneal laparoscopic para-aortic lymphadenectomy; Retroperitoneal laparoscopic aortic lymphadenectomy; Retroperitoneal laparoscopic para-aortic lymphadenectomy
  Arms: Extraperitoneal

SUMMARY:
The purpose of this study is to determine whether the extraperitoneal approach is better than the transperitoneal approach for laparoscopic aortic lymphadenectomy for the surgical staging of endometrial or ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of endometrial cancer confirmed by histopathological analysis (endometrial biopsy) requiring surgical staging according to FIGO (the International Federation of Gynecology and Obstetrics) recommendations
* Diagnosis of ovarian cancer confirmed by histopathological analysis after an initial cystectomy or oophorectomy without suspicion of neoplasia thus requiring additional surgical staging according to FIGO recommendations

Exclusion Criteria:

* Diagnosis of advanced endometrial cancer based on findings on imaging techniques (CT, MRI and/or PET)
* Diagnosis of advanced endometrial or ovarian cancer based on intraoperative findings (e.g. peritoneal carcinomatosis at initial laparoscopy)
* Patients who underwent previous aortic lymphadenectomy
* Patients who received previous pelvic and/or aortic radiotherapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2014-07 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of lymph nodes | After aortic lymphadenectomy is completed
  The number of lymph nodes (absolute number) is specified by the pathologist on histopathological analysis of the sample sent by the surgeon after surgical staging is realized (laparoscopic aortic lymphadenectomy). This variable is subdivided into: supra-mesenteric and infra-mesenteric.

SECONDARY OUTCOMES:
Operative time | At the time of the surgery
  Total duration of surgery (from initial skin incision to end of skin suture), and total aortic lymphadenectomy time (time spent since the beginning of aortic lymphadenectomy to its completion). Metric: minutes.
Intraoperative complications | At the time of surgery
  Number of patients presenting intraoperative complications. This variable is also classified according to the type of adverse outcome.
Early Postoperative complications | within 30 days after surgery
  Number of patients presenting postoperative complications. This variable is also classified according to the type of adverse outcome.
Late Postoperative complications | past 30 days after surgery
  Number of patients presenting postoperative complications. This variable is also classified according to the type of adverse outcome.
Overall survival | up to 3 years
  Number of patients alive after surgery.
Disease-free survival | up to 3 years
  Metric: months. Period of time in which there is no appearance of the symptoms or effects of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gil Moreno, M.D., PhD, Study Chair — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona; Berta Díaz Feijoo, M.D., PhD, Study Director — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona; Jose Luis Sánchez, M.D., Principal Investigator — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona; Alejandro Correa Paris, M.D., Principal Investigator — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona; M. Assumpció Pérez-Benavente, M.D., PhD, Principal Investigator — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona; Silvia Cabrera Díaz, M.D., Principal Investigator — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona; Silvia Franco Camps, M.D., Principal Investigator — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona; Oriol Puig Puig, M.D., Principal Investigator — Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona
Locations (1):
- Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona, Bacelona, Barcelona, Spain

REFERENCES:
- [Background] Gil-Moreno A, Franco-Camps S, Cabrera S, Perez-Benavente A, Martinez-Gomez X, Garcia A, Xercavins J. Pretherapeutic extraperitoneal laparoscopic staging of bulky or locally advanced cervical cancer. Ann Surg Oncol. 2011 Feb;18(2):482-9. doi: 10.1245/s10434-010-1320-9. Epub 2010 Sep 14. PMID 20839058
- [Background] Gil-Moreno A, Diaz-Feijoo B, Perez-Benavente A, del Campo JM, Xercavins J, Martinez-Palones JM. Impact of extraperitoneal lymphadenectomy on treatment and survival in patients with locally advanced cervical cancer. Gynecol Oncol. 2008 Sep;110(3 Suppl 2):S33-5. doi: 10.1016/j.ygyno.2008.03.024. Epub 2008 Jun 5. PMID 18538379
- [Background] Gil-Moreno A, Maffuz A, Diaz-Feijoo B, Puig O, Martinez-Palones JM, Perez A, Garcia A, Xercavins J. Modified approach for extraperitoneal laparoscopic staging for locally advanced cervical cancer. J Exp Clin Cancer Res. 2007 Dec;26(4):451-8. PMID 18365538
- [Background] Gil-Moreno A, Diaz-Feijoo B, Morchon S, Xercavins J. Analysis of survival after laparoscopic-assisted vaginal hysterectomy compared with the conventional abdominal approach for early-stage endometrial carcinoma: a review of the literature. J Minim Invasive Gynecol. 2006 Jan-Feb;13(1):26-35. doi: 10.1016/j.jmig.2005.08.013. PMID 16431320
- [Background] Dowdy SC, Aletti G, Cliby WA, Podratz KC, Mariani A. Extra-peritoneal laparoscopic para-aortic lymphadenectomy--a prospective cohort study of 293 patients with endometrial cancer. Gynecol Oncol. 2008 Dec;111(3):418-24. doi: 10.1016/j.ygyno.2008.08.021. Epub 2008 Oct 2. PMID 18835020
- [Background] Magrina JF, Kho R, Montero RP, Magtibay PM, Pawlina W. Robotic extraperitoneal aortic lymphadenectomy: Development of a technique. Gynecol Oncol. 2009 Apr;113(1):32-5. doi: 10.1016/j.ygyno.2008.11.038. Epub 2009 Jan 21. PMID 19157527
- [Background] Franco-Camps S, Cabrera S, Perez-Benavente A, Diaz-Feijoo B, Bradbury M, Xercavins J, Gil-Moreno A. Extraperitoneal laparoscopic approach for diagnosis and treatment of aortic lymph node recurrence in gynecologic malignancy. J Minim Invasive Gynecol. 2010 Sep-Oct;17(5):570-5. doi: 10.1016/j.jmig.2010.03.020. Epub 2010 Jun 30. PMID 20580322
- [Derived] Diaz-Feijoo B, Correa-Paris A, Perez-Benavente A, Franco-Camps S, Sanchez-Iglesias JL, Cabrera S, de la Torre J, Centeno C, Puig OP, Gil-Ibanez B, Colas E, Magrina J, Gil-Moreno A. Prospective Randomized Trial Comparing Transperitoneal Versus Extraperitoneal Laparoscopic Aortic Lymphadenectomy for Surgical Staging of Endometrial and Ovarian Cancer: The STELLA Trial. Ann Surg Oncol. 2016 Sep;23(9):2966-74. doi: 10.1245/s10434-016-5229-9. Epub 2016 Apr 20. PMID 27098143